CLINICAL TRIAL: NCT03988010
Title: Evaluation of the Effect of Preoperative Intravenous Amantadine Sulfate on the Postoperative Early Cognitive Functions in a Elderly Patient With Laparoscopic Radical Prostatectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Gülen Güler, Professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2011-KAEK-80
Record Dates: First submitted 2019-05-30; First posted 2019-06-17 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: amantadine sulphate; postoperative cognitive dysfunction; laparoscopic radical prostatectomy
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Amantadine

STUDY DESIGN:
Intervention Model Description: Patients randomly allocated to two treatment groups: Amantadine Sulphate group (Group I) and the placebo group (Group II). Participants will receive two doses of amantadine sulphate in the form of three-hour infusions. The first infusion will be administered 8 hours before the operation and the second infusion will be terminated just before the operation.
Who Masked: Participant, Care Provider
Masking Description: Randomise double blind placebo- controlled study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amantadine Sulphate (Experimental): 200 mg ıv Amantadine Sulphate in 500 cc solution
  Interventions: Drug: Amantadine Sulfate
- Placebo group (Placebo Comparator): iv 500 cc %0.9 sodium chloride
  Interventions: Drug: Placebo (for amantadine sulphate)

INTERVENTIONS:
Drug: Amantadine Sulfate — 200mg/500ml i.v. solution for infusion
  Arms: Amantadine Sulphate
Drug: Placebo (for amantadine sulphate) — 500 cc 0.9% sodium chloride
  Arms: Placebo group

SUMMARY:
Evaluation of the effect of preoperative intravenous administration of amantadine sulfate on the prevention of the development of early cognitive dysfunction in elderly patients undergoing laparoscopic radical prostatectomy

DETAILED DESCRIPTION:
Investigators believe that the preoperative prophylactic amantadine sulphate will reduce the incidence of postoperative cognitive disfunction (POCD) in patients with laparoscopic radical prostatectomy due to the neuroprotective effect, alertness enhancing effect and neuron protective effects.

ELIGIBILITY:
Inclusion Criteria:

- ASA II-III Patient

Exclusion Criteria:

* history of disease related to central nervous system, history of psychiatric disease, history of previous open heart surgery, history of previous craniotomy, renal insufficiency, hepatic failure, history of arrhythmia pre-applied standardized Mini Mental Test (sMMT) less than 24 points

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Mini Menthal Test | 24 hours after surgery
  cognitive function scale, Patients will be administered 24 hours after surgery.

SECONDARY OUTCOMES:
Verbal analog Pain Scores on rest and movement | 48 hours after surgrey
  A Research assistant, blinded to the group allocation, interviewed patients and collected data at 5 times intervals ( 2, 4, 6, 12, 24, 48 hours) in the 48 hours postoperatively. Patients were asked to rate their pain using verbal analog scale, where 0= no pain and 10= worst pain possible.

CONTACTS AND LOCATIONS:
Overall Officials: Gulen Guler, Study Director — TC Erciyes University
Locations (1):
- Erciyes Univercity, Kayseri, Melikgazi, Turkey (Türkiye)

REFERENCES:
- [Result] Moller JT, Cluitmans P, Rasmussen LS, Houx P, Rasmussen H, Canet J, Rabbitt P, Jolles J, Larsen K, Hanning CD, Langeron O, Johnson T, Lauven PM, Kristensen PA, Biedler A, van Beem H, Fraidakis O, Silverstein JH, Beneken JE, Gravenstein JS. Long-term postoperative cognitive dysfunction in the elderly ISPOCD1 study. ISPOCD investigators. International Study of Post-Operative Cognitive Dysfunction. Lancet. 1998 Mar 21;351(9106):857-61. doi: 10.1016/s0140-6736(97)07382-0. PMID 9525362
- [Result] Rasmussen LS, Johnson T, Kuipers HM, Kristensen D, Siersma VD, Vila P, Jolles J, Papaioannou A, Abildstrom H, Silverstein JH, Bonal JA, Raeder J, Nielsen IK, Korttila K, Munoz L, Dodds C, Hanning CD, Moller JT; ISPOCD2(International Study of Postoperative Cognitive Dysfunction) Investigators. Does anaesthesia cause postoperative cognitive dysfunction? A randomised study of regional versus general anaesthesia in 438 elderly patients. Acta Anaesthesiol Scand. 2003 Mar;47(3):260-6. doi: 10.1034/j.1399-6576.2003.00057.x. PMID 12648190
- [Result] Zhang J, Tan H, Jiang W, Zuo Z. Amantadine alleviates postoperative cognitive dysfunction possibly by increasing glial cell line-derived neurotrophic factor in rats. Anesthesiology. 2014 Oct;121(4):773-85. doi: 10.1097/ALN.0000000000000352. PMID 25251457
- [Result] Saletu B, Anderer P, Semlitsch HV, Grunberger J, Linzmayer L, Chaudhry HR. Amantadine infusions in mild dementia: acute double-blind placebo-controlled EEG mapping and psychometric studies. Arch Gerontol Geriatr. 1992 Jul-Aug;15(1):43-58. doi: 10.1016/0167-4943(92)90039-7. PMID 15374380